CLINICAL TRIAL: NCT04852302
Title: Managing Cancer and Living Meaningfully (CALM) Therapy in Individuals Diagnosed With a Primary Central Nervous System Tumor
Brief Title: Managing Cancer and Living Meaningfully (CALM) Therapy in Individuals Diagnosed With a Primary Brain Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Camphausen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000293; 000293-C
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: Psychological Distress; Cancer; psychotherapy; virtual therapy; Telehealth
MeSH Terms: conditions — Depression; Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy (Experimental): Remote Cancer and Living Meaningfully (CALM) therapy for participants with newly or recurrent PCNST
  Interventions: Behavioral: Cancer and Living Meaningfully (CALM) Therapy

INTERVENTIONS:
Behavioral: Cancer and Living Meaningfully (CALM) Therapy — The Cancer and Living Meaningfully (CALM) intervention is a brief, individualized psychotherapeutic intervention established to meet an unmet need to address psychological distress and promote well-being in advanced cancer patients.

SUMMARY:
Background:

Psychological distress affects many people diagnosed with a primary central nervous system tumor (CNST). Distress can include negative feelings such as anger, fear, or sadness. Researchers want to see if a type of therapy called Cancer and Living Meaningfully (CALM) can help. It promotes well-being in people who have cancer that cannot be cured.

Objective:

To find out if the CALM therapy can help people with a CNST suffering from distress.

Eligibility:

English-speaking adults ages 18 and older who have a CNST and are taking part in NIH protocol #16C0151.

Design:

This study will not take place in person. It will be done by smartphone, computer, or tablet.

Participants will fill out 7 surveys. The surveys will take 40 to 60 minutes to complete. They are all electronic. They will ask about physical and emotional symptoms, depression, feelings about death and dying, feelings about close relationships, and general well-being.

Participants will be assigned to a CALM therapist. They will have 3 to 6 individual therapy sessions in 6 months. Each session will last 45 to 60 minutes. Sessions may be audio recorded. If needed, participants may have extra sessions.

CALM includes symptom management and discussions of meaning, purpose, and mortality.

Participants may have a family member take part in at least one CALM session with them.

After the third CALM session, participants will be asked questions about CALM.

After 3 and 6 months, participants will complete the 7 surveys again.

Participation will last about 6 months.

DETAILED DESCRIPTION:
Background:

* Psychological distress is an emotional state experienced by primary central nervous system tumor (PCNST) patients throughout the illness trajectory. It can often be under identified in this patient population.
* Limited therapeutic interventions in managing distress symptoms can allow symptoms to linger without tailored mechanisms to manage the emotional challenges experienced with a tumor diagnosis. Individualized therapy in advanced cancer patients is a preferred method over pharmacological interventions when managing psychological distress, but more evidence-based research is needed to address the benefits.
* The Cancer and Living Meaningfully (CALM) intervention is a brief, individualized psychotherapeutic intervention established to meet an unmet need to address psychological distress and promote well-being in advanced cancer patients. Previous studies implementing the CALM intervention have focused on metastatic and advanced cancer patients and have reported positive effects. Implementing the CALM intervention in a sample of PCNST patients will be one of the first studies to identify the preliminary effectiveness.

Objective:

-To demonstrate the effects of the CALM intervention in reduction of depressive symptoms using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression scale in PCNST participants, from baseline to 6 months.

Eligibility:

* Adult participants greater than or equal to 18 years of age with a PCNST diagnosis who are undergoing standard of care or experimental treatment.
* The ability of the subject to speak English
* Subjects who have a life expectancy of at least 3 months from time of study entry to allow for participation in the 3 required sessions.
* The ability of the subject to understand and willing to sign a written informed consent document as determined by the assessment of the clinical team.

Design:

* A total of 100 participants will be enrolled
* Neuro-Oncology participants being seen in the clinical center or receiving telehealth services will be screened to participate. Participants will be assigned a CALM therapist, and all sessions will be completed remotely.

Data from standardized measures will be collected at 3 timepoints (Baseline, 3 months, 6 months) and qualitative interviews will be completed after the 3rd CALM session for a select number of participants until data saturation is reached (estimated to be 15-30).

-Approximate time for sessions is 45-60 minutes.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects with histological or imaging confirmation of primary central nervous system tumor (PCNST) who are undergoing standard of care or experimental treatment.
* Adults (greater than or equal to 18 years of age) who are English-speaking
* Subjects who have a life expectancy of at least 3 months from time of study entry to allow for participation in the 3 required sessions.
* Subjects must be enrolled on the Neuro-Oncology Branch Natural History Study 16C0151.
* The ability of the subject to understand and the willingness to sign a written informed consent document as determined by the assessment of the treating physicians.

EXCLUSION CRITERIA:

-Participants without access to a smartphone, computer, or tablet to complete remote sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. All collected individual participant data (IPD) will be available after primary analysis have been published.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Acquaye-Mallory A, Rodin G, Managoli M, Robins KR, Stockdill ML, Leeper HE, Vera E, Mendoza T, King AL, Cassidy ML, Gilbert MR, Armstrong TS. Managing Cancer and Living Meaningfully Therapy Delivered as a novel remote intervention in individuals diagnosed with a Primary Central Nervous System Tumor. medRxiv [Preprint]. 2026 Jan 8:2026.01.07.26343618. doi: 10.64898/2026.01.07.26343618. PMID 41542659
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000293-C.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Started | 19
Completed | 15
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Did not complete CALM therapy. | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.53 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Change of Depressive Symptoms Using the Patient-Reported Outcomes Measurement Information System (PROMIS) -Depression Scale in Primary Central Nervous System Tumor (PCNST) Participants
Description: To demonstrate the effects of the Cancer and Living Meaningfully (CALM) Therapy intervention in change of depressive symptoms using the Patient-Reported Outcomes Measurement Information System (PROMIS) -Depression scale in primary central nervous system tumor (PCNST) participants, from baseline to 6 months using a paired t-test from baseline to 6 months at a 5% significance level. PROMIS is an 8-item assessment that measures depressive symptoms within the past 7 days and participants rank symptoms on a scale that includes never, rarely, sometimes, often and always. T-scores range from 0 to 100 with T-score greater than 60 indicating moderate-severe depression.
Time Frame: Baseline to 6 months
Population: 15/19 participants completed the study and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 15
T-score
  Baseline | 54.79 (8.78)
  6 Months | 52.98 (9.88)
  Overall mean difference in change in PROMIS-Depression score from baseline to 6 months | 1.81 (1.1)
Statistical Analysis 1: Comparison: Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy; Null hypothesis was that the mean difference between the paired observations is zero; Test type: Equivalence — We evaluated the same group to determine whether their reported depression was the same, worse, or better at 6-months compared to baseline; p = 0.168, paired sample t-Test, 2-sided — The a priori threshold for statistical significance was < 0.05. We did not adjust for multiple comparisons as this was exploratory; Mean Difference (Net) = -1.81, 95% CI 2-sided [-4.47 to 0.86], Standard Deviation 4.81

2. Secondary Outcome: Mean Difference in Change of Depressive Symptoms Using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression Scale in Primary Central Nervous System Tumor (PCNST) Participants
Description: To demonstrate the short-term effects of the Cancer and Living Meaningfully (CALM) Therapy intervention in change of depressive symptoms using the Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression scale in primary central nervous system tumor (PCNST) participants from baseline to 3 months using a paired t-test from baseline to 6 months at a 5% significance level. PROMIS is an 8-item assessment that measures depressive symptoms within the past 7 days and participants rank symptoms on a scale that includes never, rarely, sometimes, often and always. T-scores range from 0 to 100 with T-score greater than 60 indicating moderate-severe depression.
Time Frame: Baseline compared at 3 months
Population: 15/19 participants completed the study and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 15
T-score
  Baseline | 54.79 (8.78)
  3 Months | 54.49 (9.85)
  Overall mean difference in change in Depressive Symptoms score from baseline to 3 months | 0.3 (1.07)
Statistical Analysis 1: Comparison: Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy; Test type: Equivalence — We evaluated the same group to determine whether their reported depression was the same, worse, or better at 3-months compared to baseline; p = 0.752, paired sample t-Test, 2-sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.30, 95% CI 2-sided [-2.29 to 1.69], Standard Deviation 3.59

3. Secondary Outcome: Change of Anxiety Score Using the Death and Dying Distress Scale (DADDS)
Description: To determine the effects of the Cancer and Living Meaningfully (CALM) Therapy intervention on death anxiety at both 3 and 6 months, compared to baseline. Total scores, subscale scores, and/or t-scores (if applicable) were completed at baseline, month 3 and month 6 and summarized, using a paired t-test from baseline to 6 months at a 5% significance level. The DADDS uses a 15-item scale to measure death anxiety. Scores range from 0-75 and higher scores mean greater distress.
Time Frame: 3 and 6 months compared to baseline
Population: 15/19 participants completed the study and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 15
Score on a scale
  Baseline | 29 (15)
  3 Months | 25 (19)
  6 Months | 27 (19)
  Overall change in Anxiety score from baseline to 3 months | 4 (4)
  Overall change in Anxiety score from baseline to 6 months | 2 (4)
Statistical Analysis 1: Comparison: Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy; Test type: Equivalence — We evaluated the same group to determine whether their reported anxiety via the Death and Dying Distress Scale was the same, worse, or better at 3-months compared to baseline; p = 0.285, paired sample t-Test, 2-sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -4.67, 95% CI 2-sided [-13.67 to 4.34], Standard Deviation 16.26
Statistical Analysis 2: Comparison: Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy; Test type: Equivalence — We evaluated the same group to determine whether their reported anxiety via the Death and Dying Distress Scale was the same, worse, or better at 6-months compared to baseline; p = 0.628, paired sample t-Test, 2-sided — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.20, 95% CI 2-sided [-11.74 to 7.34], Standard Deviation 17.22

4. Secondary Outcome: Number of Participants in a Primary Central Nervous System Tumor (PCNST) Population Eligible for Remote Cancer and Living Meaningfully (CALM) Therapy
Description: Here are the number of participants with a primary central nervous system tumor (PCNST) eligible for remote Cancer and Living Meaningfully (CALM) Therapy.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 19
Participants | 19

5. Secondary Outcome: Mean Accrual Rate for a Proportion of Participants With a Primary Central Nervous System Tumor (PCNST) Participants Per Month Using Remote Cancer and Living Meaningfully (CALM) Therapy
Description: Mean accrual rate was assessed from baseline to 6 months.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: proportion of participants per month
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 19
proportion of participants per month | 0.49 [0.27 to 0.71]

6. Secondary Outcome: Proportion of Participants Diagnosed With a Primary Central Nervous System Tumor (PCNST) Who Are Compliant Assessed by Remote Cancer and Living Meaningfully (CALM) Therapy
Description: Compliance is defined as at least 80% of participants completing the outcome measures (e.g., depression, distress, quality of life) at all time points - baseline to 6 months.
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 19
proportion of participants
  Baseline | 1 [0.55 to 1.45]
  6 Months | 0.79 [0.39 to 1.19]

7. Secondary Outcome: Serious and/or Non-serious Adverse Events in a Primary Central Nervous System Tumor (PCNST) Population Using Remote Cancer and Living Meaningfully (CALM) Therapy
Description: Here is the number of participants with a primary central nervous system tumor (PCNST) who experienced serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0) assessed from baseline to 6 months. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 19
Participants
  Baseline | 0
  6 Months | 0

8. Secondary Outcome: Proportion of Participants With a Primary Central Nervous System Tumor (PCNST) Who Participated in Remote Cancer and Living Meaningfully (CALM) Therapy and Completed the Study
Description: Here is the proportion of participants who participated in the Remote Cancer and Living Meaningfully (CALM) Therapy and completed the study
Time Frame: Baseline to 6 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 19
Proportion of participants
  Baseline | 1 [0.55 to 1.45]
  6 Months | 0.79 [0.39 to 1.19]

9. Secondary Outcome: Participant Satisfaction in a Primary Central Nervous System Tumor (PCNST) Population Using Remote Cancer and Living Meaningfully (CALM) Therapy
Description: Participant satisfaction was measured using the Was It Worth It (WIWI) questionnaire, which is designed to measure a participant's opinion of their participation. WIWI questions are dichotomous (yes/no) and are tailored to be specific to the intervention involved in the study. For the purposes of this study, there were four yes/no questions that ascertain the participants' satisfaction with the CALM intervention.
Time Frame: Baseline to 6 months
Population: 14/19 participants were analyzed because 2 did not complete CALM, 2 withdrew from the study and 1 participant did not fill out the satisfaction form.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 14
Participants
  Participants reported they would participate in the CALM intervention again. | 11
  Participants reported their quality of life changed by participating in the CALM intervention. | 10
  Participants reported that the CALM intervention was worthwhile. | 14
  Participants reported that they would recommend the CALM intervention to others with their illness | 14

10. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From the first study intervention, baseline evaluations through study participation, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
Number analyzed (Participants) | 19
Participants | 0

ADVERSE EVENTS:
Time Frame: From the first study intervention, baseline evaluations through study participation, up to 6 months.
Arm/Group | Arm 1/Remote Cancer and Living Meaningfully (CALM) Therapy
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT04852302/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT04852302/ICF_001.pdf